CLINICAL TRIAL: NCT02550158
Title: A Randomized Controlled Study Evaluating the Impact of an Educational Program "EDU-MICI" on Patients With Inflammatory Bowel Disease
Brief Title: A Study Evaluating the Impact of an Educational Program (EDU-MICI) on Patients With Inflammatory Bowel Disease
Acronym: ECIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: GETAID 2009-1
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's Disease; Ulcerative Colitis; Educational program; Inflammatory Bowel Disease; Psycho-pedagogic score; IBD
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educated Group (Experimental): Training of patients by the educational program "EDU-MICI"
  Interventions: Procedure: Educational program EDU-MICI
- Control group (Other): During the first 6 months : no training of patients by the educational program "EDU-MICI". Then, a crossover allowed uneducated patients to benefit from the educational program the next 6 months.
  Interventions: Procedure: Educational program EDU-MICI

INTERVENTIONS:
Procedure: Educational program EDU-MICI

SUMMARY:
This study has the objective to demonstrate that an education program could have a significant impact on Inflammatory Bowel Disease (IBD) patient's skills with regards to their disease.

ELIGIBILITY:
Inclusion Criteria

* Male or female patients 18 -70 years of age
* Recent diagnosis (less than 6 months) of Crohn's Disease or ulcerative colitis OR patients with an oldest pathology with a new flare, a complication and / or need to optimize medical therapy

Exclusion Criteria

* Patients unable to understand and follow the program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Psycho-pedagogic score (ECIPE score) | 6 months after Inclusion
  Variation of a psycho-pedagogic score (ECIPE score) measured at baseline and 6 months after inclusion.

SECONDARY OUTCOMES:
Hospitalization | 6 months after inclusion
  Number of hospitalizations >24h
Disease Flare | 6 months after inclusion
  Number of disease flare
Major complication | 6 months after inclusion
  Number of major complication = number of serious adverse events related to the disease
Quality of life | 6 months after inclusion
  Variation of score for the Simple Inflammatory Bowel Disease Questionnaire (SIBDQ)
Observance | 6 months after inclusion
  Variation of score for the "Observance" questionnaire
Patient concerns | 6 months after inclusion
  Variation of score for the "Rating Form of Inflammatory Bowel Disease Patient Concerns" (RFIPC) questionnaire.
Work productivity | 6 months after inclusion
  Variation of score for the "Work Productivity and Activity Impairment - General Health" (WPAI-GH) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Allez, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Jacques Moreau, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (18):
- France (18):
  - Chu Amiens, Amiens
  - Hopital Beaujon, Clichy
  - Hopital Louis Mourier, Colombes
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - Hopital Nord, Marseille
  - Chi Le Raincy Montfermeil, Montfermeil
  - Chu Montpellier, Montpellier
  - Chu Nantes, Nantes
  - CHU NICE, Nice
  - Hopital Saint Louis, Paris
  - Hopital Saint-Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - Chu Rouen, Rouen
  - Chu Saint-Etienne, Saint-Priest-en-Jarez
  - Chu Toulouse, Toulouse
  - Hopital Tourcoing, Tourcoing
  - Chu Tours, Tours

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- See also: Related Info — http://www.getaid.org